CLINICAL TRIAL: NCT06068543
Title: A Phase 2 Randomized Controlled Trial of Epigallocatechin-3-Gallate (EGCG) on Frailty and Inflammation in Older Survivors of Cancer
Brief Title: Reducing Frailty for Older Cancer Survivors Using Supplements II
Acronym: ReFOCUS2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Nikesha Gilmore, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UOCPC23048
Record Dates: First submitted 2023-09-20; First posted 2023-10-05 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Frailty; Inflammation
MeSH Terms: conditions — Frailty; Inflammation | interventions — epigallocatechin gallate; microcrystalline cellulose; Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Patients in the intervention Arm will receive 800 mg Epigallocatechin-3-Gallate (EGCG) + 250mg Ascorbic Acid
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Epigallocatechin-3-Gallate (EGCG) (Experimental): 800mg Epigallocatechin-3-Gallate (EGCG) pills AND 250mg Ascorbic Acid (Vitamin C) once daily
  Interventions: Drug: Epigallocatechin-3-Gallate (EGCG); Dietary Supplement: Ascorbic Acid (Vitamin C)
- Microcrystalline cellulose (MCC) (Placebo Comparator): 800mg microcrystalline cellulose (MCC) pills AND 250mg Ascorbic Acid (Vitamin C) once daily
  Interventions: Drug: Microcrystalline cellulose (MCC); Dietary Supplement: Ascorbic Acid (Vitamin C)

INTERVENTIONS:
Drug: Epigallocatechin-3-Gallate (EGCG) — 800mg Epigallocatechin-3-Gallate (EGCG)
  Other Names: EGCG
  Arms: Epigallocatechin-3-Gallate (EGCG)
Drug: Microcrystalline cellulose (MCC) — 800mg microcrystalline cellulose (MCC)
  Other Names: MCC
  Arms: Microcrystalline cellulose (MCC)
Dietary Supplement: Ascorbic Acid (Vitamin C) — 250mg Ascorbic Acid (Vitamin C) taken one time daily for 12 weeks
  Other Names: Vitamin C

SUMMARY:
This study is a two-arm placebo controlled randomized clinical trial, to assess the effect of a 12-week EGCG intervention on physical frailty compared to placebo in pre-frail older cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

1. Be age 65 or over.
2. Be diagnosed with stage I-III Cancer
3. Have completed curative intent treatment ≤10 years prior to screening Patients on the following endocrine therapies are allowed to enroll (Anastrozole,Leuprolide acetate, and Bicalutamide)
4. Have a Fried's Frailty Score (FFS) of ≥ 1
5. Able to provide informed consent

Exclusion Criteria:

1. Have chemotherapy or other systemic cancer treatment planned to occur during the study period.
2. Have abnormal liver function tests (ALT, AST, and bilirubin) per most recent available lab test (within 3 months of screening)

   * 3 times institutional upper limit of normal for ALT and AST
   * 1.5 times institutional upper limit of normal for bilirubin
3. Have uncontrolled or unmanaged liver disease.
4. Consume more than 6 cups of green tea per day.
5. Have known allergies to caffeine.
6. Be diagnosed with a major psychiatric illness requiring hospitalization within the last year.
7. Be diagnosed with dementia.
8. Cannot provide informed consent due to lack of decision-making capacity (as determined by the patient's oncologist).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of physical frailty measured using the Short Physical Performance Battery (SPPB) in patients in the EGCG arm compared to placebo; change in SPPB scores from baseline to 12 weeks. | 12 Weeks
  We will assess the change in SPPB scores from baseline to 12 weeks after baseline in patients in the EGCG intervention arm compared to the placebo arm.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States